CLINICAL TRIAL: NCT03710265
Title: A Phase I, Open-label Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of SHR-1701 in Subjects With Metastatic or Locally Advanced Solid Tumors and Expansion to Selected Indications
Brief Title: SHR-1701 in Metastatic or Locally Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-I-101
Record Dates: First submitted 2018-10-14; First posted 2018-10-18 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Solid Tumor
Keywords: SHR-1701; Solid tumor; Metastatic or locally advanced solid tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1701 (Experimental)
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — Subjects will receive an intravenous infusion of SHR-1701 in a dose escalation until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.

SUMMARY:
The main purpose of this Phase I study is to access the safety and tolerability of SHR-1701 at different dose levels. It is hoped to find out the recommended dose for Phase II/III.

DETAILED DESCRIPTION:
This is a Phase I, open-label trial in patients with metastatic or locally advanced solid tumor. There are three parts of the study: a dose-escalation part, a dose-expansion part, and a clinical expansion part. Dose escalation part is a standard "3+3" cohort design, for which 3 or 6 subjects will be enrolled at each dose level depending on the occurrence of dose-limiting toxicities (DLTs). Dose-expansion means that at least 10 subjects (included subjects of the dose-escalation part) will be selected in 2 - 3 dose levels to focus on the pharmacokinetics (PK) / pharmacodynamic (PD) features. After determination of the recommended dose for Phase II (RP2D), clinical expansion will be opened. Many more subjects will be invited to take part in the study and received the study drug at the RP2D. Additional purpose of the study is to find out whether the study drug has anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 75 years
* Life expectancy >= 12 weeks as judged by the Investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Has measurable disease per RECIST 1.1
* Subjects with confirmed metastatic or locally advanced solid tumor (histologically or cytologically) and there is no known effective anti-tumor treatment (refractory or relapsed from standard treatment).
* Adequate hematological, hepatic and renal function as defined in the protocol
* Females of childbearing potential (FOCBP), who are not surgically sterile or postmenopausal, must conduct pregnancy test (serum or urine) within 7 days before enrollment, and must not be pregnant or breast-feeding women. If the result is negative, she must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs. And non-sterilized males who are sexually active must agree to use adequate contraception during the experiment and 3 months after the last administration of the test drugs.
* Able to understand and sign an informed consent, and able to comply with all procedures

Exclusion Criteria:

* Anticancer treatment within 28 days before the first dose of study drug
* Major surgery within 28 days before start of trial treatment (prior diagnostic biopsy is permitted)
* Systemic therapy with immunosuppressive agents within 7 days prior to the first dose of study drug; or use any investigational drug within 28 days before the start of trial treatment
* With any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism, except for subjects with vitiligo or resolved childhood asthma/atopy. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded
* Subjects with active central nervous system (CNS) metastases causing clinical symptoms or metastases that require therapeutic intervention are excluded
* Clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, Congestive heart failure (New York heart association (NYHA) class > 2), or ventricular arrhythmia which need medical intervention.
* History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy, e.g., hepatitis B or C
* Previous malignant disease (other than the target malignancy to be investigated in the trial) within the last 2 years. Subjects with history of cervical carcinoma in situ, superficial or non-invasive bladder cancer or basal cell or squamous cell cancer in situ previously treated with curative intent are NOT excluded.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability profile of SHR-1701 | Up to week 3
  Number of Subjects who occurs dose-limiting toxicity (DLTs)
Objective Response Rate (ORR) assessed by site investigator as per RECIST 1.1 | Screening up to study completion, an average of 1 year

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SHR-1701 | Up to 4 weeks after last treatment
Peak Plasma Concentration (Cmax) of SHR-1701 | Up to 4 weeks after last treatment
Half-time (t1/2) of SHR-1701 | Up to 4 weeks after last treatment
Pharmacodynamic features of SHR-1701 | 12 months (anticipated)
  SHR-1701 receptor occupation
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors | 12 months (anticipated)
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ¡Ý30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Disease Control Rate (DCR) per RECIST 1.1 | 12 months (anticipated)
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1.
Best Overall Response (BOR) per RECIST 1.1 | 12 months (anticipated)
Immunogenicity of SHR-1701 | 12 months (anticipated)
  anti SHR-1603 antibodies (ADA)
Trough plasma concentration (C trough) of SHR-1701 | Up to 4 weeks after last treatment
Immunogenicity of SHR-1701 | 12 months (anticipated)
Disease Control Rate (DCR) per RECIST 1.1 | 12 months (anticipated)
Clinical Benefit Rate(CBR) per RECIST 1.1 | 12 months (anticipated)
Progression-Free Survival (PFS) per RECIST 1.1 | 12 months (anticipated)
Duration of Response (DoR) per RECIST 1.1 | 12 months (anticipated)
Overall Survival (OS) | 12 months (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu D, Zhou J, Wang Y, Li M, Jiang H, Liu Y, Yin X, Ge M, Xiang X, Ying J, Huang J, Zhang YQ, Cheng Y, Huang Z, Yuan X, Han W, Yan D, Wang X, Liu P, Wang L, Zhang X, Luo S, Liu T, Shen L. Bifunctional anti-PD-L1/TGF-betaRII agent SHR-1701 in advanced solid tumors: a dose-escalation, dose-expansion, and clinical-expansion phase 1 trial. BMC Med. 2022 Oct 25;20(1):408. doi: 10.1186/s12916-022-02605-9. PMID 36280870